CLINICAL TRIAL: NCT00196859
Title: Ibandronate With or Without Capecitabine in Elderly Patients With Early Breast Cancer
Brief Title: Study in Elderly Patients With Early Breast Cancer (ICE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GBG Forschungs GmbH (Other)
Collaborators: Hoffmann-La Roche (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBG 32; BIG 4-04
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2011-08

CONDITIONS: Breast Cancer
Keywords: Early Breast Cancer in elderly Patients; Ibandronate plus/minus Capecitabine in elderly patients
MeSH Terms: conditions — Breast Neoplasms | interventions — Ibandronic Acid; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Ibandronate 50 mg p.o. daily or 6 mg i.v., q4W, 2yrs
  Interventions: Drug: Ibandronate
- B (Experimental): Ibandronate 50 mg p.o. daily or 6 mg i.v., q4W, 2yrs plus Capecitabine 2000 mg/m2 days 1-14 q d22 x6
  Interventions: Drug: Ibandronate, Capecitabine

INTERVENTIONS:
Drug: Ibandronate, Capecitabine — Ibandronate 50 mg p.o. daily or 6 mg i.v., q4W, 2yrs plus Capecitabine 2000 mg/m2 days 1-14 q d22 x6
  Arms: B
Drug: Ibandronate — Ibandronate 50 mg p.o. daily or 6 mg i.v., q4W, 2yrs
  Arms: A

SUMMARY:
This trial is done to determine the role of adjuvant chemotherapy with capecitabine in patients ≥ 65.

DETAILED DESCRIPTION:
Title of the study:

Ibandronate with or without Capecitabine in Elderly Patients with Early Breast Cancer - (ICE Study)

Rationale:

Approximately 50% of new diagnosis of early breast cancer is made in patients above the age of 65. As this age group has not been eligible for most trials in the past, the effect of adjuvant therapy is still unclear in elderly patients. The primary aim of this trial will be to determine the role of adjuvant chemotherapy with capecitabine in elderly patients. The high activity, acceptable toxicity and oral formulation of this compound especially meet the requirements of elderly patients.

Bisphosphonates are of established effectivity in treatment and prevention of osteoporosis. Furthermore, two studies have recently shown that adjuvant long term use of clodronate can reduce the risk of recurrence of breast cancer. The third generation bisphosphonate ibandronate will be given in this trial to all patients to prevent osteoporosis and recurrence from breast cancer, both conditions these patients are at risk. As the preference of elderly patients for intravenous or oral application is not known, the mode of application of ibandronate will be according to patients' choice and the preference and compliance will be a secondary endpoint.

Primary objective

To compare the event-free survival in elderly patients after local treatment for primary breast cancer treated with either ibandronate alone or ibandronate and capecitabine as adjuvant treatment

Secondary objectives

To compare the overall survival between the two arms

To determine the compliance in both arms

To determine the toxicity in both arms

To determine the rate of bone-related events in hormone sensitive and insensitive disease (with or without endocrine therapy)

To determine the preference to oral or intravenous application of ibandronate

To assess quality of life

To compare a geriatric assessment by Charlson versus VES 13 score

Tertiary objective

To determine prognostic factors on tumor tissue collected from primary surgery and to correlate them with study treatment effect

To evaluate the prognostic impact of age, serum albumin, hemoglobin level, creatinine clearance, Charlson Score, VES-Score in a multivariate analysis for the prediction of treatment associated adverse events and limited life time expectancy

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to beginning specific protocol procedures, including expected cooperation of the patients for the treatment and follow-up, must be obtained and documented according to the local regulatory requirements.
2. Histologically confirmed unilateral or bilateral primary carcinoma of the breast.
3. Age at diagnosis ≥ 65 years
4. Adequately surgical treatment with complete resection (Ro) of the tumor and > or = 10 axillary nodes. Sole sentinel node biopsy is allowed if the sentinel node shows no tumor involvement.
5. Node positive disease irrespective of additional risk factors or node negative disease with at least one other risk factor (histologic tumor size > or = 2 cm, grade II or III, ER and PR negative)
6. No evidence for distant metastasis after complete diagnostic work up
7. Performance Status ECOG < or = 2
8. Charlson Scale of < or = 2
9. Estimated life expectancy of at least 5 years (irrespective of breast cancer diagnosis)
10. The patient must be accessible for treatment and follow-up.

Exclusion Criteria:

1. Known hypersensitivity reaction to the compounds or incorporated substances or known dihydropyrimidine dehydrogenase deficiency.
2. Inadequate organ function including: Leucocytes < 3,5 G/l, Platelets < 100 G/l , Bilirubin 1.25 times above normal limits, Creatinine clearance calculated by the Cockroft-Gold formula of above 50 ml/min, uncompensated cardiac function, severe and relevant co-morbidity that would interact with the application of cytotoxic agents or the participation in the study
3. Another primary malignancy with an event-free survival of < 5 years, except curatively treated basalioma of the skin
4. Time since axillary dissection > 3 months
5. Locally advanced, non-operable breast cancer
6. Previous invasive breast carcinoma
7. Previous treatment with cytotoxic agents for any reason
8. Concurrent treatment with hormonal replacement therapy (treatment should be stopped before entering the trial).
9. Previous treatment with bisphosphonates for osteoporosis is allowed, however this treatment has to be substituted by the trial medication
10. Concurrent specific systemic anti-tumor treatment or treatment with experimental compounds within the last 6 months
11. Concurrent treatment with other tumor specific experimental drugs. Participation in another clinical trial with any investigational not marketed drug within 30 days prior to study entry.
12. Concurrent treatment with virostatic agents like brivudine or analoga sorivudine, concurrent treatment with aminoglycosides
13. Male patients

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2004-06; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Any local or distant relapse of breast cancer, any second malignancy, and any death irrespective of its cause

SECONDARY OUTCOMES:
Any death related and not-related to breast cancer
Any premature treatment discontinuation of capecitabine or ibandronate
Any grade II to grade IV AE specified to serious or non serious events
Every bone fracture, bone surgery, new diagnosis of osteoporosis
Completed months of i.v. or p.o. treatment with ibandronate
Frequency of changes of preference of Ibandronate application
Evaluation according to EORTC Q 30

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Nitz, MD, Principal Investigator — Evangelisches Krankenhaus Bethesda, Mönchengladbach
Locations (1):
- Prof. Dr. med. Ulrike Nitz, Mönchengladbach, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Schmidt M, Nitz U, Reimer T, Schmatloch S, Graf H, Just M, Stickeler E, Untch M, Runnebaum I, Belau A, Huober J, Jackisch C, Hofmann M, Krocker J, Nekljudova V, Loibl S; GBG/AGO-B, NOGGO/WSG study groups. Adjuvant capecitabine versus nihil in older patients with node-positive/high-risk node-negative early breast cancer receiving ibandronate - The ICE randomized clinical trial. Eur J Cancer. 2023 Nov;194:113324. doi: 10.1016/j.ejca.2023.113324. Epub 2023 Sep 7. PMID 37797387
- [Derived] Hoon SN, Lau PK, White AM, Bulsara MK, Banks PD, Redfern AD. Capecitabine for hormone receptor-positive versus hormone receptor-negative breast cancer. Cochrane Database Syst Rev. 2021 May 26;5(5):CD011220. doi: 10.1002/14651858.CD011220.pub2. PMID 34037241
- See also: Click here for more information about this study: ICE Study — http://www.germanbreastgroup.de